CLINICAL TRIAL: NCT01219972
Title: Prospective Cohort Study of Late Pulmonary Complications in Patients Who Received Allogeneic Hematopoietic Stem Cells Transplantation: Estimation of Incidence and Identification of Distinct Nosologic Entities
Brief Title: Pulmonary Complications of Allografts
Acronym: ALLOPULM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC 04118
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Pulmonary Complications
Keywords: Bone marrow transplant; Pulmonary complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allografted patients: * All consecutive patients who underwent an allogeneic blood stem cells transplantation performed at saint Louis hospital during the study recruitment period
  * if alive at 100 days post-transplant
  * and who gave informed consent

SUMMARY:
This is a prognostic study of the late lung complications arising at the patient's having received an allograft of hematopoetic stem cells.

DETAILED DESCRIPTION:
* Objectives To estimate the incidence of late (at least occurring 100 days after transplantation) pulmonary complications following allogeneic blood stem cells transplantation
* Study Design Prospective Cohort Study All follow-up data were actualiized in September, 2016.
* Sample Size 200 transplanted patients
* Main Endpoint Non infectious pulmonary complications within the first 3 years

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic Blood stem cell transplantation
* Alive at day 100 post-transplant

Exclusion Criteria:

* Non informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a allogeneic blood stem cell transplantation, alive at 100 days post-transplantation
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Non infectious pulmonary complication | 3 years

SECONDARY OUTCOMES:
Survival after non infectious pulmonary complication | 3 years and 10 years
Overall survival | 3 years and 10 years
Long term time course of Pulmonary Function Tests (PFTs) | 3 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bergeron - Laffaurie,, PhDMD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bergeron A, Chevret S, Peffault de Latour R, Chagnon K, de Margerie-Mellon C, Riviere F, Robin M, Mani J, Lorillon G, Socie G, Tazi A. Noninfectious lung complications after allogeneic haematopoietic stem cell transplantation. Eur Respir J. 2018 May 3;51(5):1702617. doi: 10.1183/13993003.02617-2017. Print 2018 May. PMID 29650555